CLINICAL TRIAL: NCT01484223
Title: Efectiveness of a Cognitive Behavioral Intervention in Patients With Symptoms Somatization, as Measure Quality of Life, Front the Clinical Practice Usual Action in Primary Health Care. A Controlled Clinical Trial With Parallel Groups
Brief Title: Effectiveness of Cognitive Behavioral Intervention in Patients With Symptoms Somatization in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gerencia de Atención Primaria, Madrid (Other Government)
Collaborators: Instituto de Salud Carlos III (Other Government); Fondo de Investigacion Sanitaria (Other)
Responsible Party: Principal Investigator, Esperanza Escortell, Epidemiologist, Gerencia de Atención Primaria, Madrid
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: FIS PI08/90707
Record Dates: First submitted 2011-11-30; First posted 2011-12-02 (Estimated); Last update posted 2012-10-11 (Estimated); Status verified 2012-10

CONDITIONS: Quality of Life
Keywords: Primary Health Care; Somatization symptoms; Cognitive Behavioral Therapy; Nursing intervention
MeSH Terms: interventions — Cognitive Behavioral Therapy; Primary Health Care; Methods; Quality of Life

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental Group (Experimental): Intervention group: Structured nursing intervention
  Interventions: Behavioral: Cognitive Behavioral Therapy
- No intervention (No Intervention): Control group: conventional intervention or non_support

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — Four Cognitive behavioral group sessions. Each session will last two hours a week
  Other Names: Primary Health Care; Somatization symptoms; Nursing intervention; Quality of life
  Arms: Experimental Group

SUMMARY:
The purpose of this study is to evaluate the efectiveness of a behavioral cognitive grupal intervention (BCI) in patients with somatization symptoms which has an effect on the perceived quality of life front conventional intervention.

DETAILED DESCRIPTION:
Aim: to determine whether a cognitive-behavioral group intervention in patients with unexplicated somatic symptoms, that have come to the primary care medical in Madrid, is more effective than normal practice in terms of improving life quality at one year.

Method:

Design:cluster randomized trial. Setting: study in Health Centers Primary Care of Area of Madrid Health Service. unit of randomization are centres.Analysis unit: patients between 18 and 65 years old.

Intervention: The cognitive behavioral grupal Terapy in the internention group and the usual intervention in the control group.

Sample size adjusted for design effect=242 (121 in each arm). Main response variable: preceived quality of life (SF-12).

Data Analysis:comparison of the proportion of patients that improve in 4 or more points in the area of Mental Healthcare from the SF-12 in both groups,at 6 months and 1 year after patient inclusion.

ELIGIBILITY:
Inclusion Criteria:

* Attending patients with 2 or more medically unexplained somatic symptoms during the last 6 months.
* Having came to medical examination on primary care at least 10 times during the last year.
* be able to follow the trial´s demands, not have plans for moving another place and understand the Spanish language.
* Patients who consent to take part.

Exclusion Criteria:

* Diagnostics on serious mental disorder.
* Suicidal intentions at the moment of getting involved in the study.
* Diagnostics on addiction to toxic substances.
* Diagnostics on well-known body illness responsible for the symptoms.
* Previous psychotherapy during the previous year.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2009-10; Primary Completion 2012-04 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Perceived quality of life | Change from baseline in quality of life at 12 months after the intervention
  Perceived quality of life: Quality of life measured by SF-12 questionnare on Mental Healthcare Change from baseline in quality of life at 3, 6 and 12 months after the intervention.

SECONDARY OUTCOMES:
Questionnarie on Global Clinical Impression | Change from baseline in patient and doctor´s perception at 12 months afer the intervention
  It is used to assess the patient´s(PGI questionnarie) and the doctor´s(CGI questionnarie)perception on the former´s improvement after the interventions have been carried out. It will be undertaken 6 and 12 moths later, so as to assess the effectiveness of the group intervention.
Number of examinations | Number of examinations from baseline until 12 months after the intervention
  Number of requested and programmed doctor´s examinations during the period of study (itemized between infirmary and medicine)
Prescribed medicine | Prescribed medicine from baseline until 12 months after the intervention
  Prescribed medicine during the period of study, with doubtful therapeutic value for their processing, related to the unexplained somatic symptoms. The included medicines are those related to the functional symptomatology
Temporary labor disability (TLD) | Days on TLD from baseline until 12 months after the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Alberto López García-Franco, MD, Principal Investigator — Gerencia Atención Primaria. Madrid
Locations (1):
- Gerencia Atención Primaria, Madrid., Madrid, Madrid, Spain

REFERENCES:
- [Derived] Lopez-Garcia-Franco A, del-Cura-Gonzalez MI, Caballero-Martinez L, Sanz-Cuesta T, Diaz-Garcia MI, Rodriguez-Monje MT, Chahua M, Munoz-Sanchez I, Serrano-Gonzalez D, Rollan-Llanderas T, Nieto-Blanco E, Losada-Cucco L, Caballero-Martinez F, Sanz-Garcia N, Pose-Garcia B, Jurado-Sueiro M, Rey ML, de Blas Gonzalez FG, Abanto MA, Bayona TS, Ayllon-Camargo R, Lopez IS, Hernando ML, Beltran-Alvarez R, Aguilar-Gutierrez AI, Mota-Rodriguez JL, Cosculluela-Pueyo R, Lopez-Martin-Aragon T, Bonilla-Sanchez R, Aritieda-Gonzalez-Granda MC, Razola-Rincon R, Sanchez-de-la-Ventana MA, Martinez-Guinea C, Huerta-Galindo L, Barrio-Ovalle AB, Miguel-Martin S, Portero-Fraile P, Pensado-Freire H, Herrera-Garcia ML, Azcoaga-Lorenzo A, Gomez-Garcia I, Llamas-Sandino N, Lopez-Borja I, Maldonado-Castro H, Lumbreras-Villaran P, Ascanio-Duran C. Effectiveness of a cognitive behavioral intervention in patients with medically unexplained symptoms: cluster randomized trial. BMC Fam Pract. 2012 May 2;13:35. doi: 10.1186/1471-2296-13-35. PMID 22551252